CLINICAL TRIAL: NCT05670431
Title: The Effect of Smile Designs Using the Digital Smile Design Program on Aesthetic Perception
Brief Title: The Effect of Smile Designs on Aesthetic Perception
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Aysegul Kurt, Associate Professor, Trakya University
Other Study IDs: TUTF-GOBAEK 2021/534
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-04

CONDITIONS: Dentistry; Perception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 4th-grade students of a dentistry faculty
- 5th-grade students of a dentistry faculty
- Dentists
- Specialist dentists
- Laypeople

SUMMARY:
The goal of this observational study is to examine the effect of designs using different aesthetic dental proportions made with the digital smile design program on the aesthetic perception of individuals of different ages, gender, and educational status.

The main questions it aims to answer are:

1. The golden ratio is the most aesthetic ratio known and accepted in dentofacial structures.
2. There is no significant difference between the aesthetic perception of dental students, dentists, specialist dentists and laypeople.

Participants will answer:

* The first 5 questions related that demographic data such as age, gender, and educational status.
* The smile designs of a woman and a man, prepared according to 8 different principles, will be evaluated by the participants according to the Likert scale.

Researchers will compare the 4th and 5th-grade students of a dentistry faculty, dentists, specialist dentists and laypeople to see the effect of smile design on facial aesthetic perception.

ELIGIBILITY:
Inclusion Criteria:

* Anyone who can answer the survey online

Exclusion Criteria:

* individuals under the age of 18

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 4th and 5th-grade students of a dentistry faculty: 4th and 5th-grade students at the university where the researcher works (Trakya University, Faculty of Dentistry)
  Dentists and specialist dentists: Dentists and specialist dentists working in health institutions in the country where the researcher is located (Republic of Türkiye)
  Laypeople: People who came to the dental faculty for treatment, relatives and friends of the researcher.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Likert scale | 1 day (single measurement)
  There are 5 rating levels on the Likerts scale: very ugly, ugly, unstable, beautiful, very beautiful. People in 5 different groups will evaluate different smile designs with a Likert scale according to their aesthetic perceptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Merkez, Edirne, Turkey (Türkiye)